CLINICAL TRIAL: NCT07374445
Title: The Timing for Liraglutide in Patients Remaining Obese at 6 Months After Metabolic Surgery: an Observational Study
Brief Title: Research on Timing of Liraglutide Therapy in Patients With Obesity After Metabolic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-507-02
Record Dates: First submitted 2025-09-01; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Weight Loss; Bariatric Surgery
Keywords: Liraglutide; bariatric surgery; obesity; BMI; GLP-1 receptor agonists
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Liraglutide; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Sham Comparator): Receive guidance on diet and exercise throughout the program, without the use of drugs
  Interventions: Behavioral: Diet and exercise guidelines
- Liraglutide 6 month group (Experimental): Receive guidance on diet and exercise throughout the program, started pharmacological intervention at enrollment for 6 months.
  Interventions: Drug: Liraglutide injection; Behavioral: Diet and exercise guidelines
- Liraglutide 9 month group (Experimental): Receive guidance on diet and exercise throughout the program, started pharmacological intervention 6 months post 3 months of enrollment.
  Interventions: Drug: Liraglutide injection; Behavioral: Diet and exercise guidelines
- Liraglutide 12 month group (Experimental): Receive guidance on diet and exercise throughout the program, started pharmacological intervention 6 months post 6 months of enrollment.
  Interventions: Drug: Liraglutide injection; Behavioral: Diet and exercise guidelines

INTERVENTIONS:
Drug: Liraglutide injection — Patients received a 24-week regimen of once-daily liraglutide, initiated at 0.6 mg/day and titrated weekly by 0.6 mg to a maximum tolerated dose of up to 3.0 mg/day.
  Arms: Liraglutide 12 month group; Liraglutide 6 month group; Liraglutide 9 month group
Behavioral: Diet and exercise guidelines — Participants followed a science-based diet and exercise program intervention

SUMMARY:
The goal of this clinical trial is to compare the weight loss and metabolic benefit in patients remaining obesity at 6 months after metabolic surgery. The main questions it aims to answer are:

[primary hypothesis 1] Whether liraglutide benefits weight loss when it is initiated early after metabolic surgery.

[primary hypothesis 2] Whether weight loss and metabolic benefits are greater when linaglutide is initiated in patients who are obese at 6 months after metabolic surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients 6 months after metabolic surgery;
* 18 years ≤ age ≤ 65 years;
* Body Mass Index (BMI) ≥ 28 kg/m^2

Exclusion Criteria:

* allergy to liraglutide, severe hepatic or renal impairment (eGFR <60 mL/min/1.73 m² or ALT/AST ≥3× ULN)
* history of medullary thyroid carcinoma, MEN-2 or other malignancies
* pancreatitis or severe gastrointestinal disease, pregnancy or lactation
* use of anti-obesity drugs or other interventional trials within 3 months or major uncontrolled illness
* Patients were discontinued if withdrawn, intolerant, lost to follow-up, or developed severe adverse events.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in %TWL from baseline to endpoint across patient groups | 48 weeks from enrollment
  %TWL = ([baseline weight - weight at follow-up]/baseline weight) × 100%. The measurement of body weight is in kilograms. %TWL represents the percentage of total weight loss, measured in percent.
  This indicator reflects the percentage of weight loss from the baseline.
  The mean and standard deviation of %TWL were calculated for subjects within each group. Subsequently, intergroup comparisons were performed to calculate p-values. If p < 0.05, pairwise comparisons were further conducted. Based on the final results, the differences in weight loss among groups were evaluated.

SECONDARY OUTCOMES:
Change in BMI from baseline to endpoint across patient groups | 48 weeks from enrollment
  BMI = Weight / Height^2 weight and height will be combined to report BMI in kg/m^2 (Weight is measured in kilograms, height in meters, and BMI is expressed in kilograms per square meter) The observed metric is the difference obtained by subtracting the endpoint BMI from the baseline BMI.
  Complete data correction for each patient using baseline values, then calculate overall mean and SD by group. Subsequently perform intergroup comparisons to compute P-values; if P < 0.05, proceed with pairwise comparisons.
Change in body composition from baseline to endpoint across patient groups | 48 weeks from enrollment
  body composition (Including body fat, fat-free mass, skeletal muscle, etc.; in kilograms） Body composition values at the endpoint minus baseline values are used as the change metric to evaluate body composition changes (These indicators are used to assess the body composition improvement of patients)
  Complete data correction for each patient using baseline values, then calculate overall mean and SD by group. Subsequently perform intergroup comparisons to compute P-values; if P < 0.05, proceed with pairwise comparisons.
Changes in blood pressure from baseline to endpoint | 48 weeks from enrollment
  Difference between the endpoint blood pressure and the baseline value.(blood pressure in mmHg; This indicator is used to assess improvements in a patient's blood pressure.) Complete data correction for each patient using baseline values, then calculate overall mean and SD by group. Subsequently perform intergroup comparisons to compute P-values; if P < 0.05, proceed with pairwise comparisons.
Changes in fasting blood glucose from baseline to endpoint | 48 weeks from enrollment
  Difference between endpoint fasting blood glucose and baseline value (blood glucose in mmol/L; This indicator is used to assess improvements in patients' fasting blood glucose levels.) Complete data correction for each patient using baseline values, then calculate overall mean and SD by group. Subsequently perform intergroup comparisons to compute P-values; if P < 0.05, proceed with pairwise comparisons.
Change in HbA1c from baseline to endpoint across patient groups | 48 weeks from enrollment
  Difference between the endpoint HbA1c value and the baseline value (HbA1c in percentage, This indicator is used to assess improvements in a patient's HbA1c levels.) Complete data correction for each patient using baseline values, then calculate overall mean and SD by group. Subsequently perform intergroup comparisons to compute P-values; if P < 0.05, proceed with pairwise comparisons.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No
No participant data are available